CLINICAL TRIAL: NCT01168323
Title: Spaced Education to Optimize Prostate Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard University Faculty of Medicine (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); American Urological Association (Other); Astellas Pharma US, Inc. (Industry); National Institutes of Health (NIH) (NIH); Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: B. Price Kerfoot MD EdM, Harvard Medical School; Veterans Affairs Boston Healthcare System.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: M15310; IRB# 1786 (Other: Veterans Affairs Boston Healthcare System); 5K08HS017147 (AHRQ)
Record Dates: First submitted 2010-07-20; First posted 2010-07-23 (Estimated); Last update posted 2010-08-09 (Estimated); Status verified 2010-07

CONDITIONS: Prostate Cancer
Keywords: Medical Education; Educational Technology; Clinical Practice Guideline; Prostate specific antigen
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spaced education clinicians - cohort 1 (Experimental): Spaced education clinicians receive four isomorphic cycles of 9 spaced education emails over 36-weeks (0-2 emails per week). Each email contained one question-explanation.
  Interventions: Behavioral: Online spaced education
- Control clinicians - cohort 2 (No Intervention): Control clinicians received no intervention

INTERVENTIONS:
Behavioral: Online spaced education — Spaced education is currently delivered via periodic emails that contain clinical case scenarios and multiple-choice questions. Upon submitting answers to each question online, clinicians receive immediate feedback and educational material. The questions are then repeated over spaced intervals of time to harness the pedagogical benefits of the spacing effect.
  Arms: Spaced education clinicians - cohort 1

SUMMARY:
Two memory research findings (the spacing and testing effects) can dramatically improve retention of learning, but they have largely have been ignored by educators. The researchers have developed a novel form of online education (termed 'spaced education') based on these two effects which has been shown in randomized trials to improve knowledge acquisition and boost learning retention. Using prostate cancer screening as an experimental system, the researchers investigated whether spaced education could durably improve clinicians' behaviors, not just their knowledge.

ELIGIBILITY:
Inclusion Criteria:

* Primary care providers (physicians, nurse practitioners, and physician assistants) from the 8 Veterans Affairs (VA) hospitals in the New England region (Veterans Integrated Service Network 1 [VISN-1]) were eligible to enroll.

Exclusion Criteria:

* Primary care providers (PCPs) who ordered PSA as a screen for prostate cancer less than 10 times each year were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2007-01; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Percentage of inappropriate prostate-specific antigen (PSA) screening performed by clinicians | Weeks 1-108
  The primary outcome measure was the difference in the percentage of inappropriate PSA screening performed by clinicians in the spaced education and control cohorts. Based on published clinical guidelines and reports, inappropriate PSA utilization was defined as the use of PSA for prostate cancer screening in patients >76 or <40 years old, or with an estimated life expectancy of less than 10 years.

SECONDARY OUTCOMES:
Change in test scores between cohorts measured in weeks 1-36 | Weeks 1-36
Change in spaced education performance measured in weeks 1-36 | Weeks 1-36
Clinicians' intention to participate in future spaced education programs | Week 36
  Assessed on end-of program survey at week 36
Time required by clinicians to complete the spaced education questions-explanations | Week 36
  Assessed on end-of program survey at week 36

CONTACTS AND LOCATIONS:
Overall Officials: B. Price Kerfoot, MD EdM, Principal Investigator — VA Boston Healthcare System, Harvard Medical School
Locations (1):
- Veterans Affairs Boston Healthcare System, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Kerfoot BP, Lawler EV, Sokolovskaya G, Gagnon D, Conlin PR. Durable improvements in prostate cancer screening from online spaced education a randomized controlled trial. Am J Prev Med. 2010 Nov;39(5):472-8. doi: 10.1016/j.amepre.2010.07.016. PMID 20965387